CLINICAL TRIAL: NCT01399931
Title: Dual Point Acquisition in the Interim Pet Scan Performed During ABVD Treatment, in Early-Stage Hodgkin's Lymphoma Patients With Bulky Lesions
Brief Title: Dual Point PET Scan in Early Stage Hodgkin Lymphoma Patients With Bulky Lesions
Acronym: 2P-HD-10
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Santa Croce-Carle Cuneo (Other)
Collaborators: Consorzio Mario Negri Sud (Other); Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Principal Investigator, DR. ANDREA GALLAMINI, HEAD OF HAEMATOLOGY DEPT. A.S.O. S. CROCE AND CARLE, Ospedale Santa Croce-Carle Cuneo
Other Study IDs: 2P-HD-10 STUDY
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Hodgkin's Lymphoma
Keywords: Early stage
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Early-stage Hodgkin Lymphoma Patients: Early-stage Hodgkin Lymphoma (HL) patients presenting bulky nodal lesions treated with ABVD and consolidation radiotherapy

SUMMARY:
To assess specificity and overall accuracy of interim dual-point acquisition PET in predicting treatment outcome.

The study is aimed at assessing the specificity of interim dual-point PET performed after 2 ABVD cycles to predict treatment outcome in early-stage Hodgkin's Lymphoma patients presenting bulky lesions at baseline.

DETAILED DESCRIPTION:
The proposed study is an non-interventional survey of a cohort of patients in whom interim PET scan is performed only for prognostic aims.

PET with 18F-FDG is a standard staging procedure for most lymphoma subtypes. Performed early during the therapy for Hodgkin's lymphoma (HL) its results have a high prognostic value and is the main predictor of treatment outcome. From 2006 onward, interim-PET after 2 ABVD courses has been increasingly performed in the daily clinical practice as a routine test for disease prognosis, and now it can be considered as a standard prognostic tool.

The novelty of the study relies on a new method for interim-PET scan execution: a dynamic study, with 2 different time points of image acquisition. This could potentially enable us to discriminate between unspecific, inflammatory DG uptake, from a "true" uptake form persisting viable neoplastic cells. Therefore, the main aim of the study is reducing false positive results in the interim-PET scan interpretation. Since dynamic changes of FDG uptake in Hodgkin's lymphoma are still unknown we propose, in the present study, to assess the by the same acquisition technique the pattern of FDG uptake at baseline in untreated patients affected by this neoplasm.

The Institutions equipped with a Magnetic Resonance scanners and a diffusion weighted imaging analysis technique (DW-MRI), could participate to the DW-MRI sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Hodgkin lymphoma diagnosis according all the WHO classification subtype but lymphocyte predominance.
* Age 18 - 60 years old
* stage IA- IIA (by FDG-PET scan)
* Presence of bulky tumour (either in Mediastinum or other site)
* Treatment with ABVD x 4 (early stage)
* Consolidation Radiotherapy on bulky lesion
* Signed the Informed consent form

Exclusion Criteria:

* Diabetes mellitus uncompensated
* Lymphocyte predominance histology
* Pregnancy or lactation
* Implanted biomedical devices (for DW-MRI sub study)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Early-stage Hodgkin Lymphoma (HL) patients presenting bulky nodal lesions.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-10 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Event free survival (EFS) | 1 year
  To assess feasibility of using interim dual-point acquisition PET in real world of clinical practice as well as describing the outcome of early stage HL patients.

SECONDARY OUTCOMES:
Evaluation of inflammation markers prognostic role | 3 years
  To assess prognostic value of inflammation markers (ESR, CRP, Ferritin, Transferrin, Fibrinogen, Alpha 2-globulins) as biomarkers of treatment outcome in early stage HL patients

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Gallamini, MD, Principal Investigator — Azienda Sanitaria Ospedaliera Santa Croce e Carle Cuneo
Locations (6):
- Italy (6):
  - Ospedale Santi Antonio E Biagio E Cesare Arrigo, Alessandria, AL
  - Azienda Sanitaria Ospedaliera S. Croce E Carle, Cuneo, Cuneo
  - Azienda Ospedaliera Universitaria S. Martino, Genova, GE
  - Azienda Ospedaliera S. Gerardo, Monza, MB
  - Azienda Ospedaliera Ospedali Riuniti Papardo Piemonte, Messina, ME
  - Azienda Ospedaliera S. Giovanni Battista, Torino, TO

REFERENCES:
- [Background] Gallamini A.:Positron emission tomography scanning: a new paradigm for the management of Hodgkin's lymphoma. Haematologica 2010;95, 1-3 Gallamini A, Rigacci L, Merli F, Nassi L, Bosi A, Capodanno I, et al. The predictive value of positron emission tomography scanning performed after two courses of standard therapy on treatment outcome in advanced stage Hodgkin's disease. Haematologica 2006 Apr;91(4):475-81. Meignan M, Itti E, Gallamini A, Haioun C. Interim 18F-fluorodeoxyglucose positron emission tomography in diffuse large B-cell lymphoma: qualitative or quantitative interpretation - where do we stand? Leukemia & Lymphoma 2009; 50(11) 1753-56. Gallamini A, Hutchings M, Rigacci L, Specht L, Merli F, Hansen M, et al. Early interim 2-[18F]fluoro-2-deoxy-D-glucose positron emission tomography is prognostically superior to international prognostic score in advanced-stage Hodgkin's lymphoma: a report from a joint Italian-Danish study. J Clin Oncol 2007 Aug 20;25(24):3746-52.